CLINICAL TRIAL: NCT04703075
Title: Safety and Tolerability of Ultra-short Course Rifapentine and Isoniazid (1HP) for Prevention of Tuberculosis in HIV-Uninfected Individuals
Brief Title: Ultra Curto (Ultra Short) TB Prevention Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00284317; U01AI152961 (NIH)
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine; Isoniazid

STUDY DESIGN:
Intervention Model Description: Arm A (n=250): Experimental arm. Rifapentine 600 mg daily and isoniazid 300 mg daily for 4 weeks.
  Arm B (n=250): Control arm. Rifapentine 900 mg and isoniazid 900 mg weekly for 12 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: 1HP (Experimental): Participants will receive Rifapentine 600 mg daily and isoniazid (INH) 300 mg daily for 4 weeks.
  Interventions: Drug: Rifapentine 600 mg and INH 300 mg
- Arm B: 3HP (Active Comparator): Participants will receive Rifapentine 900 mg and isoniazid 900 mg weekly for 12 weeks.
  Interventions: Drug: Rifapentine 900 mg and INH 900 mg

INTERVENTIONS:
Drug: Rifapentine 600 mg and INH 300 mg — Participants will receive Rifapentine 600 mg and INH 300 mg
  Arms: Arm A: 1HP
Drug: Rifapentine 900 mg and INH 900 mg — Participants will receive Rifapentine 900 mg and INH 900mg
  Arms: Arm B: 3HP

SUMMARY:
To compare treatment success (adherence and completion of treatment) and safety of 1HP with 3HP in HIV-uninfected adults and adolescents at increased risk of TB.

DETAILED DESCRIPTION:
Tuberculosis (TB) is the leading infectious killer globally and a major cause of illness and suffering. The World Health Organization has prioritized TB preventive therapy (TPT) for people with latent TB infection (LTBI) as a key strategy for controlling the epidemic. Prevention of TB with isoniazid preventive therapy (IPT) is effective and reduces morbidity and mortality, and has been the mainstay of TB prevention for decades. But for an intervention with an excellent evidence of efficacy, global uptake has been abysmal. Completion rates for IPT when it is administered are poor (Gillespie 2008; Durovni 2010), with a large proportion of patients unable to complete treatment (McClintock 2017; Sterling 2011). While uptake is influenced by a variety of factors, a critical element has been the duration of IPT, with adherence falling sharply over time in clinical trials and practice. Shorter course regimens have a much higher completion rate and are more acceptable to patients, clinicians, and programs.

ELIGIBILITY:
Inclusion Criteria:

* Positive tuberculin skin test or interferon-gamma release assay (IGRA) test and
* Household contact of an infectious TB case within previous 90 days, defined as sleeping at least once in a residence with a person diagnosed with pulmonary TB, or
* Documented conversion of Tuberculin skin test (TST)/IGRA from negative to positive within 2 years

Exclusion Criteria:

* Documented HIV infection
* Evidence of active tuberculosis on clinical exam or chest x-ray
* Known intolerance of any study drug
* Treatment for active or latent TB in the past for more than 14 days
* Known close contact to someone with INH or rifampin resistant TB
* Active liver disease or Aspartate aminotransferase(AST)/Alanine transaminase (ALT) >3 times upper limit of normal (ULN)
* Neutropenia (ANC <1000)
* Peripheral neuropathy >Grade 1 by DAIDS Grading Table
* Pregnant or breastfeeding. Women of childbearing potential must agree to use non-hormonal contraception during study treatment.
* Weight <40 kg

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Chaisson, MD, Principal Investigator — Johns Hopkins University
Locations (2):
- Brazil (2):
  - Fundacao de Medicina Tropical Doutor Heitor, Manaus, Amazonas
  - NAPDOT, Rio de Janeiro, Rio de Janeiro

REFERENCES:
- [Derived] Durovni B, Cordeiro-Santos M, Cavalcante SC, Spener-Gomes R, Garcia J, Cohn S, Saraceni V, Kohler B, Moulton LH, Brito da Souza A, Berihun A, Marzinke M, Chaisson RE; Ultra Curto Study Team. Acceptability and safety of one versus three months of rifapentine and isoniazid to prevent tuberculosis in people exposed in the household or workplace in Brazil: The Ultra-Curto randomized controlled trial. PLoS Med. 2026 Feb 10;23(2):e1004758. doi: 10.1371/journal.pmed.1004758. eCollection 2026 Feb. PMID 41666121

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 531 people signed consent to be screened for eligibility. 31 people did not meet the eligibility criteria. The reasons were: Risk for Bad Outcome n=8, Active TB n=5, Withdrew Consent n=3, Pregnant n=1, Neutropenia n=2, AST/ALT > 3 times ULN n=8, HIV infection n= 1, Drug-Drug Interaction n=2, Past TB-TPT treatment n=1. 500 people were assigned to a treatment group in the study. 249 were Randomized to Arm A:1HP. 251 were randomized to Arm B: 3HP
Period: Overall Study
Arm/Group | Arm A: 1HP | Arm B: 3HP
Started | 249 | 251
Completed | 223 | 211
Not Completed | 26 | 40
Not completed — Adverse Event | 11 | 7
Not completed — Lost to Follow-up | 6 | 12
Not completed — Physician Decision | 3 | 0
Not completed — Moved | 0 | 2
Not completed — Index INH Resistant | 0 | 1
Not completed — Lack of Efficacy | 6 | 18

BASELINE CHARACTERISTICS:
Population: Thirty one participants were not eligible and not randomized to the arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: 1HP | Arm B: 3HP | Total
Number analyzed (Participants) | 249 | 251 | 500
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [15 to 90] | 38 [15 to 81] | 39 [15 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 167 | 140 | 307
  Male | 82 | 111 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 23 | 61
  White | 70 | 70 | 140
  More than one race | 141 | 155 | 296
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 249 | 251 | 500

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Treatment With >90% Adherence
Description: To compare treatment success (completion of treatment with >90% adherence) of 1HP with 3HP in HIV-uninfected adults and adolescents at increased risk of TB.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 1HP | Arm B: 3HP
Number analyzed (Participants) | 249 | 251
Participants | 223 | 211
Statistical Analysis 1: Comparison: Arm A: 1HP vs Arm B: 3HP; Test type: Superiority; p = 0.07, Chi-squared, Corrected; Risk Difference (RD) = 5.5

2. Primary Outcome: Frequency of Targeted Adverse Events or Treatment Discontinuation for Side Effects
Description: Participants with targeted adverse event grade 2 or more or discontinuing treatment for any side effect.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: 1HP | Arm B: 3HP
Number analyzed (Participants) | 249 | 251
Participants | 40 | 26

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Targeted adverse events
Arm/Group | Arm A: 1HP | Arm B: 3HP
All-Cause Mortality (participants affected / at risk) | 0/249 | 0/251
Serious Adverse Events (participants affected / at risk) | 1/249 | 2/251
Other Adverse Events (participants affected / at risk) | 13/249 | 10/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 1HP (N=249) | Arm B: 3HP (N=251)
Hospitalization (Surgical and medical procedures) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: 1HP (N=249) | Arm B: 3HP (N=251)
Hepatotoxicity (Hepatobiliary disorders) | 13 (13) | 10 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04703075/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/75/NCT04703075/SAP_001.pdf